CLINICAL TRIAL: NCT03424928
Title: A Pilot, Open-label, Randomized, Two-Way Crossover, Single-Dose Bioequivalence Study of Pomalidomide Under Fasting Condition in Chinese Healthy Volunteers.
Brief Title: A Pilot Bioequivalence Study of Pomalidomide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XS-2017-001-SXYK
Record Dates: First submitted 2017-12-14; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Bioequivalence
Keywords: Pomalidomide; Multiple myeloma; Bioequivalence
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Intervention Model Description: two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomalidomide 4 MG Oral Capsule (Experimental): per os,capsule,4mg,1 capsule per period
  Interventions: Drug: Pomalidomide 4 MG Oral Capsule
- Pomalidomide 4 MG Oral Capsule-Pomalyst (Experimental): per os,capsule,4mg,1 capsule per period
  Interventions: Drug: Pomalidomide 4 MG Oral Capsule-Pomalyst

INTERVENTIONS:
Drug: Pomalidomide 4 MG Oral Capsule — per os,capsule,4mg,1 capsule per period
  Arms: Pomalidomide 4 MG Oral Capsule
Drug: Pomalidomide 4 MG Oral Capsule-Pomalyst — per os,capsule,4mg,1 capsule per period
  Arms: Pomalidomide 4 MG Oral Capsule-Pomalyst

SUMMARY:
Pomalidomide capsule were developed to offer an alternative to the marketed formulation, This pilot study was aim to pre-assess the bioequivalence of the capsule formulations under fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should read, sign and date an Informed Consent Form and be fully informed of possible adverse events prior to any study procedures.
* Subjects should complete the trial according to the regulations.
* Subjects must agree to take effective contraceptive methods to prevent pregnancy from 2 weeks before screening until 3 months of last dose administration. Subjects must agree to avoid semen and blood donation until 3 months of last dose administration.
* Healthy male volunteers of 18-50 years old.
* Body mass index (BMI) ranges from 18.0 to 28.0 kg/m2, body weight ≥ 50 kg.
* Medically healthy subjects with clinically normal Neutrophils and Platelets within 14 days.
* No history of heart, liver, kidney, gastrointestinal tract diseases, nervous system, neural abnormities or metabolic abnormalities.

Exclusion Criteria:

* Smokers (>3 cigarettes/day)
* History of allergic reactions to pomalidomide or Thalidomide analogues. Any food allergies, which in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* Any history of thrombus or liver, kidney diseases.
* History of Alcohol abuse (3990 ml beer, 1400 ml wine, 350 ml spirits/week)
* Recent donation of plasma or significant loss of whole blood (>400 ml) within 3 months.
* Subjects have difficulty to swallow or any clinical significant history of ongoing gastrointestinal problems which affect absorption of drugs.
* Received a prescription medicine within 2 weeks prior to study dosing.
* Received a non-prescription drugs, traditional Chinese medicine, health products within prior to study dosing.
* Received a special food (dragon fruit, grapefruit or other tropical fruit) or strenuous exercise within 1 week prior to study dosing. Regular use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to study administration.
* Any anticipation in other trial within 3 months.
* Abnormal laboratory tests judged clinically significant.
* Positive test result for HBsAg, HBeAg, HBeAb, HBcAB, HCvAB, HIV antibody, Syphilis screening antibody.
* Received a caffeine/Xanthine beverages or food within 48 h prior to study dosing.
* Received an alcohol within 24 h prior to study dosing or positive test result for alcohol screening.
* Positive test result for drugs of abuse.
* Other reasons which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day 1, Day 2, Day 3 of cycle 1, Day 8, Day 9, Day 10 of cycle 2.
  90% CI of T/R within 80-125%
Area under the plasma concentration versus time curve from 0 to the last measurable concentration (AUC0-t) | Day 1, Day 2, Day 3 of cycle 1, Day 8, Day 9, Day 10 of cycle 2.
  90% CI of T/R within 80-125%
Area under the plasma concentration versus time curve from 0 to infinity (AUC0-inf) | Day 1, Day 2, Day 3 of cycle 1, Day 8, Day 9, Day 10 of cycle 2.
  90% CI of T/R within 80-125%

CONTACTS AND LOCATIONS:
Overall Officials: Ruigang Hou, Bachelor, Principal Investigator — Second Hospital of Shanxi Medical University; Linhua Linhua, PhD, Principal Investigator — Second Hospital of Shanxi Medical University
Locations (1):
- The second hospital of shanxi medical university, Taiyuan, Shanxi, China